CLINICAL TRIAL: NCT00306592
Title: An Open-Label, Multicenter, Extension Study to Evaluate the Safety and Tolerability of Natalizumab Following Re-Initiation of Dosing in Multiple Sclerosis Subjects Who Have Completed Study C-1801, C-1802, or C-1803 and a Dosing Suspension Safety Evaluation
Brief Title: Natalizumab Re-Initiation of Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-MS-322
Record Dates: First submitted 2006-01-31; First posted 2006-03-24 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Experimental): All study participants in 101-MS-322 (NCT00306592) and 101-MS-321 (NCT00297232) received open label 300 mg intravenous (IV) natalizumab 60-minute infusion once every 4 weeks (28 days ±7 days) for up to 48 weeks. After 48 weeks, participants from 101-MS-322 (NCT00306592) entering study 101-MS-321 (NCT 00297232; considered the Long-Term Treatment Period of 101-MS-322) were continued on treatment from Week 52 through Week 480.
  Interventions: Biological: BG00002 (natalizumab)

INTERVENTIONS:
Biological: BG00002 (natalizumab)
  Other Names: Tysabri

SUMMARY:
The primary objectives of this study are to further evaluate the safety of natalizumab (Tysabri®) monotherapy by evaluating the risk of hypersensitivity and immunogenicity following re-exposure to natalizumab, and to confirm the safety of switching to natalizumab from interferon beta (IFN-β), glatiramer acetate (GA), or other multiple sclerosis (MS) therapies.

DETAILED DESCRIPTION:
Study 101-MS-322 (NCT00306592) is conducted to evaluate the safety of natalizumab monotherapy following re-exposure to natalizumab of former clinical trial participants in Studies C-1801 (NCT00027300), C-1802 (NCT00030966), and C-1803 (NCT00097760). This study includes participants in North America. In parallel with the conduct of this study, a similar study, 101-MS-321 (NCT00297232) is initiated for participants in Europe and the rest of the world. The primary purpose and primary outcome for both studies are identical, therefore, the combined Week 48 data from both studies are presented. In addition, after 48 weeks, participants from 101-MS-322 (NCT00306592) can enter study 101-MS-321 (NCT 00297232), which is considered the Long-Term Treatment Period of 101-MS-322 (NCT00306592).

ELIGIBILITY:
Inclusion Criteria:

* MS subjects who completed Study C-1801 (NCT00027300), C-1802 (NCT00030966), or C-1803 (NCT00097760) and completed a Dosing Suspension Safety Evaluation (neurological examination and magnetic resonance imaging [MRI] scan)
* Considered by the investigator to be free of signs and symptoms suggestive of progressive multifocal leukoencephalopathy (PML) based on medical history, physical examination, or laboratory testing (results from the Dosing Suspension Safety Evaluation from Study C-1808 [NCT000276172] may be used)
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Considered by the investigator to be immunocompromised, based on medical history, physical examination, or laboratory testing (results from the Dosing Suspension Safety Evaluation from Study C-1808 may be used), or due to prior immunosuppressive treatment
* History of persistent anti-natalizumab antibodies, based upon testing from prior natalizumab studies
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (59):
- United States (49):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Berkeley, California
  - Research Site, Los Angeles, California
  - Research Site, Redwood City, California
  - Research Site, Sacramento, California
  - Research Site, San Francisco, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Arlington, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Northbrook, Illinois
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Worcester, Massachusetts
  - Research Site, East Lansing, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Teaneck, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Syracuse, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Milwaukee, Wisconsin
- Canada (10):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Center, New York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec

REFERENCES:
- [Background] O'Connor P, Goodman A, Kappos L, Lublin F, Polman C, Rudick RA, Hauswirth K, Cristiano LM, Forrestal F, Duda P. Long-term safety and effectiveness of natalizumab redosing and treatment in the STRATA MS Study. Neurology. 2014 Jul 1;83(1):78-86. doi: 10.1212/WNL.0000000000000541. Epub 2014 Jun 4. PMID 24898925
- See also: The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families, and healthcare providers.) — http://www.nationalmssociety.org
- See also: (MSActiveSource.com is a resource for news, information, and disease management for all individuals touched by Multiple Sclerosis. This site is sponsored by Biogen Idec.) — http://www.msactivesource.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from studies 101-MS-321 (NCT00297232) and 101-MS-322 (NCT00306592) are included in this presentation of combined Week 48 data.
Groups:
- Natalizumab Study 101-MS-322 (NCT00306592): Open label 300 mg intravenous (IV) natalizumab 60-minute infusion once every 4 weeks (28 days ±7 days) for up to 48 weeks. After 48 weeks, participants from 101-MS-322 (NCT00306592) entering study 101-MS-321 (NCT00297232; considered the Long-Term Treatment Period of 101-MS-322) were continued on treatment from Week 52 through Week 480.
- Natalizumab Study 101-MS-321 (NCT00297232): Open label 300 mg intravenous (IV) natalizumab 60-minute infusion once every 4 weeks (28 days ±7 days) for up to 268 weeks. (Week 52 through Week 480 of Study 101-MS-321 (NCT00297232) is considered to be the Long-Term Treatment Period).
Period: Overall Study
Arm/Group | Natalizumab Study 101-MS-322 (NCT00306592) | Natalizumab Study 101-MS-321 (NCT00297232)
Started | 404 | 690
Completed at 24 Weeks | 207 | 0
Completed Between 24 and 48 Weeks | 85 | 0
Completed at 48 Weeks | 81 | 632
Entered 101-MS-321 Extension Study | 22 | 0 (pertains to participants transitioning from 101-MS-322 (NCT00306592) study only)
Completed | 373 | 632
Not Completed | 31 | 58
Not completed — Adverse Event | 8 | 15
Not completed — Lost to Follow-up | 1 | 0
Not completed — Noncompliance | 0 | 2
Not completed — Persistent Antibodies | 6 | 3
Not completed — Voluntary | 10 | 6
Not completed — Other | 5 | 10
Not completed — Other | 1 | 2
Not completed — 48-week Treatment Period Ongoing | 0 | 20

BASELINE CHARACTERISTICS:
Population: Participants from 101-MS-322 (NCT00306592) and 101-MS-321 (NCT00297232) are combined.
Groups:
- 300 mg Natalizumab IV Monthly: All study participants in 101-MS-322 (NCT00306592) and 101-MS-321 (NCT00297232) received open label 300 mg intravenous (IV) natalizumab 60-minute infusion once every 4 weeks (28 days ±7 days) for up to 48 weeks. After 48 weeks, participants from 101-MS-322 (NCT00306592) entering study 101-MS-321 (NCT 00297232; considered the Long-Term Treatment Period of 101-MS-322) were continued on treatment from Week 52 through Week 480.
Arm/Group | 300 mg Natalizumab IV Monthly
Number analyzed (Participants) | 1094
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (8.12)
Age, Customized [Number; unit: participants]
  ≥ 18 to < 20 years | 0
  ≥ 20 to < 30 years | 98
  ≥ 30 to < 40 years | 347
  ≥ 40 to < 50 years | 454
  ≥ 50 to < 59 years | 195
  >/= 60 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 755
  Male | 339

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: AEs: any sign, symptom, or diagnosis/disease that is unfavorable or unintended, that is new, or if pre-existing, worsens in participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. SAEs: an event that results in death; an event that, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); an outcome that results in a congenital anomaly/birth defect diagnosed in a child of a participant; an event that requires or prolongs inpatient hospitalization; an event that results in persistent or significant disability/incapacity. Any other medically important event that, in the opinion of the investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. Treatment-emergent AEs: events in participants who had received at least 1 dose of study drug, regardless of relationship to study drug.
Time Frame: Baseline through Week 48
Population: Participants receiving at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | 300 mg Natalizumab IV Monthly
Number analyzed (Participants) | 1094
participants
  AE | 826
  Moderate or severe AE | 487
  Severe AE | 66
  AE related to study drug | 161
  SAE | 61
  SAE related to study drug | 5
  Discontinuation of study drug due to AE | 24
  Withdrawal from study due to AE | 24

2. Primary Outcome: Number of Participants With Hypersensitivity-related Adverse Events
Description: For purposes of this analysis, the terms 'hypersensitivity' and 'drug hypersensitivity' were categorized by their temporal relationship to study drug infusion (within 2 hours of the start of the infusion), and were considered equivalent. Hypersensitivity reactions are defined as infusion reactions with the following preferred terms: hypersensitivity not otherwise specified (NOS), anaphylactic reaction, anaphylactoid reaction, dermatitis allergic, drug hypersensitivity, urticaria NOS, vasoconstriction, urticaria generalised, hypersensitivity, urticaria.
Time Frame: Baseline through Week 48
Population: Participants receiving at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | 300 mg Natalizumab IV Monthly
Number analyzed (Participants) | 1094
participants | 8

3. Primary Outcome: Number of Participants With Antibodies to Natalizumab
Description: 'Positive with unknown persistence' is defined as a positive result (≥0.5 micrograms/mL) at one timepoint only with no confirmatory re-test available at least 42 days later. 'Transient positive' is defined as a positive at one timepoint but negative upon re-test at least 42 days later. 'Persistent positive' is defined as positive at 2 or more timepoints separated by at least 42 days. The threshold for classifying a sample as 'antibody positive' was set at the lowest level of reactivity that had a measurable impact on drug serum concentrations.
Time Frame: Baseline (Week 0), Week 4, Week 24 (test was repeated after 8 weeks if positive, to confirm persistence)
Population: All participants who received at least 1 dose of natalizumab, had a negative baseline antibody result, and had at least 1 antibody result after the first dose.
Measure: Number; unit: participants
Arm/Group | 300 mg Natalizumab IV Monthly
Number analyzed (Participants) | 1043
participants
  Antibody negative | 1004
  Antibody positive with unknown persistence | 15
  Antibody transient positive | 8
  Antibody persistent positive | 16

ADVERSE EVENTS:
Time Frame: SAEs were collected from the time of enrollment, and AEs from the time of first dose of natalizumab, until Week 48.
Description: Participants from studies 101-MS-321 (NCT00297232) and 101-MS-322 (NCT00306592) are included in this presentation of combined Week 48 data.
Arm/Group | 300 mg Natalizumab IV Monthly
Serious Adverse Events (participants affected / at risk) | 61/1094
Other Adverse Events (participants affected / at risk) | 492/1094
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Natalizumab IV Monthly (N=1094)
Multiple sclerosis relapse (Nervous system disorders) | 21
Urinary tract infection (Infections and infestations) | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hypersensitivity (Immune system disorders) | 2
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Viral meningitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Staphyloccal infection (Infections and infestations) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaphylactic reaction (Immune system disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial fibrosis (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Small intestine obstruction (Gastrointestinal disorders) | 1
Cholecystitis (Gastrointestinal disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1
Ovarian torsion (Reproductive system and breast disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 mg Natalizumab IV Monthly (N=1094)
Multiple sclerosis relapse (Nervous system disorders) | 156
Nasopharyngitis (Infections and infestations) | 141
Upper respiratory tract infection (Infections and infestations) | 119
Headache (Nervous system disorders) | 91
Urinary tract infection (Infections and infestations) | 85
Fatigue (General disorders) | 81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.